CLINICAL TRIAL: NCT03121040
Title: Improved ATP Generation Efficiency for Younger Athletes by Ingestion of a Vespa Amino Acid Mixture
Brief Title: Clinical Trial for Vespa Amino Acid Mixture (VAAM®)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Meiji Health Science and Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 0002
Record Dates: First submitted 2017-04-01; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Sports Injury
Keywords: Vespa amino acid mixture (VAAM®); Young athletes; Nutrition; lactic acid accumulation; Anaerobic metabolism; ATP; Sports damage
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Subjects ingested VAAM® for 10 weeks (Experimental): Ten young athletes ingested Vespa amino acid mixture (VAAM®) for 10 weeks, divided into different meter race including 1500-, 800- and 400-meter races.
  Interventions: Dietary Supplement: Vespa amino acid mixture
- Subjects ingested VAAM® for 6 weeks (Experimental): Ten young athletes ingested Vespa amino acid mixture (VAAM®) for 6 weeks, divided into different meter race including 1500-, 800- and 400-meter races.
  Interventions: Dietary Supplement: Vespa amino acid mixture
- Subjects ingested nothing (No Intervention): Ten young athletes before ingesting Vespa amino acid mixture (VAAM®) , divided into different meter race including 1500-, 800- and 400-meter races.

INTERVENTIONS:
Dietary Supplement: Vespa amino acid mixture — 17 kinds of amino acids mixture in specific proportion
  Other Names: VAAM®
  Arms: Subjects ingested VAAM® for 10 weeks; Subjects ingested VAAM® for 6 weeks

SUMMARY:
ATP is generated mainly through anaerobic metabolism during strenuous exercise, which is then followed by the generation of lactic acid. However, this process can only be maintained for a short time, approximately one minute, because the accumulation of lactic acid in the muscles may affect muscle performance. The efficiency of lactic acid metabolism is one of the most important reasons for endurance improvement. The purpose of this study was to evaluate the impacts of the daily ingestion of a commercially available Vespa amino acid mixture (VAAM®) beverage on blood parameters that are related to fatigue, muscle damage and immunity in healthy, young athletes during middle-distance running exercises. VAAM® contains 17 types of amino acids at a certain ratio, and evaluations were completed during 10 weeks of consecutive required speed and strength running tests.

DETAILED DESCRIPTION:
The subjects were instructed to maintain their usual dietary habits in addition to drinking VAAM® (two cans every day) for 10 weeks. In detail, on the 6 days/week of supervised running tests, participants were instructed to consume one drink before their warm-up exercise and the other drink while running. During their sessions and without supervision (1 day/week), participants were also instructed to consume one drink in the morning after breakfast and the other drink in the evening after dinner.

The subjects were divided into three groups for the running tests: 3 males were assigned to group 1, which involved training for the 1500-meter race; 2 males were assigned to group 2, which involved training for the 800-meter race; and 1 male and 3 females were assigned to group 3, which involved training for the 400-meter race. The running exercises began with a 45 min warm-up (including jogging, leg stretching, etc.) followed by running their specific races. The experimental procedure was conducted 6 days/week for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Athletes from 16 to 18 years old;
* Subjects underwent a physical examination before enrollment and showed no sign of illness or malaise.

Exclusion Criteria:

* Subjects were smokers or ergogenic aid users;
* Subjects had any metabolic, cardiovascular, renal, or liver diseases;
* Subjects had psychiatric disorders.

Ages: 16 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2009-05-02 (Actual); Primary Completion 2009-07-16 (Actual); Study Completion 2009-07-22 (Actual)

PRIMARY OUTCOMES:
change of running time scores at 10 weeks | 10 weeks
change of the plasma lactic acid clearance rate after running at 10 weeks | 10 weeks
change of red blood cells after running at 10 weeks | 10 weeks

IPD SHARING:
Plan to Share IPD: No